CLINICAL TRIAL: NCT02661022
Title: A Phase 1/2 Open Label Study of SL-401 in Combination With Pomalidomide and Dexamethasone in Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: SL-401 in Combination With Pomalidomide and Dexamethasone in Relapsed or Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-401-0414
Record Dates: First submitted 2015-12-16; First posted 2016-01-21 (Estimated); Results first posted 2023-11-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Relapsed and Refractory; Multiple Myeloma; CD123; SL-401/pom/dex; TAG/pom/dex; R/R; MM
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1, SL-401 7 µg/kg/day (Experimental): Dose Level 1: single-agent SL-401 7 µg/kg/day on Days 1-5 during the initial 28-day run-in cycle followed by a combination of SL-401/pomalidomide/dexamethasone (pom/dex) if there was no dose-limiting toxicity during the run-in cycle
  Interventions: Drug: SL-401 7 µg/kg/day
- Phase 1, SL-401 9 µg/kg/day (Experimental): Dose Level 2: SL-401 9 µg/kg/day in combination with pom/dex
  Interventions: Drug: SL-401 9 µg/kg/day

INTERVENTIONS:
Drug: SL-401 7 µg/kg/day — SL-401 7 µg/kg/day in combination with pom/dex
  Other Names: tagraxofusp-erzs
  Arms: Phase 1, SL-401 7 µg/kg/day
Drug: SL-401 9 µg/kg/day — SL-401 9 µg/kg/day in combination with pom/dex
  Other Names: tagraxofusp-erzs
  Arms: Phase 1, SL-401 9 µg/kg/day

SUMMARY:
A Phase 1/2, Open Label Study of SL-401 in Combination with Pomalidomide and Dexamethasone In Relapsed and Refractory Multiple Myeloma

DETAILED DESCRIPTION:
This study is a phase 1/2 multicenter, open-label study of SL-401 (tagraxofusp-erzs) in combination with standard doses of pomalidomide and dexamethasone in patients with relapsed and refractory multiple myeloma (MM). The study will be conducted in 2 phases: Phase 1 is the dose-escalation phase to determine the maximum tested dose (MTD) of SL-401 in combination with standard doses of pomalidomide and dexamethasone. In Phase 1, each evaluated SL-401 dose level will incorporate an initial "Run-in Cycle" (i.e. cycle 1) of single agent SL-401 in at least 3 patients; following the Run-in Cycle, patients who have not experienced a dose-limiting toxicity (DLT) will receive combination SL-401/pomalidomide and dexamethasone in cycles 2 and beyond. All patients in Phase 2 will receive 1 cycle of SL-401 monotherapy in cycle 1, followed by combination of SL-401/pomalidomide/dexamethasone in cycle 2 and beyond. The dose of SL-401 will be the MTD of SL-401 or MTD given in combination with pomalidomide/dexamethasone determined during Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be considered for inclusion if they meet all of the following criteria. (All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrollment.)

  1. Male or female patient who is at least 18 years of age.
  2. Patient has given voluntary written informed consent before performance of any study-related procedures not part of standard (non-investigational) medical care.
  3. Patient has been previously diagnosed with MM based on standard criteria.
  4. Patient has received:

     1. At least 2 prior therapies including a proteasome inhibitor (≥ 2 cycles) and lenalidomide (≥ 2 cycles), and
     2. Has achieved at least stable disease (SD) for ≥ 1 cycle of treatment on ≥ 1 prior treatment, and
     3. Has demonstrated disease progression subsequent to treatment, during or within 90 days following completion of the most recent therapy.
  5. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2.
  6. Patient has measurable disease defined as at least 1 of the following:

     1. Serum M protein ≥ 0.5 /dL (≥5 g/L)
     2. Urine M protein ≥ 200 mg/24 hours
     3. Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
  7. Clinical Laboratory Inclusion Criteria: The following laboratory results must be met within 14 days (or as stipulated) prior to study drug (treatment) administration:

     1. Absolute neutrophil count (ANC) ≥ 1000 cells/μl (growth factor cannot be used within the previous 7 days).
     2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN).
     3. Platelet count ≥ 50,000/μl (without platelet transfusion in the previous 7 days).
     4. Total bilirubin ≤ 1.5 mg/dL.
     5. Serum creatinine ≤ 2.0 mL/dL and creatinine clearance ≥ 40 mL/min (calculated by the Cockcroft-Gault Equation or per 24 hour urine collection).
     6. Serum albumin ≥ 3.2 g/dL in the absence of receipt of (IV) albumin within the previous 72 hours.
     7. Serum creatine phosphokinase (CPK) ≤ 2.5 × the ULN.
     8. Serum calcium (corrected for albumin) level at or below the ULN range (treatment of hypercalcemia is allowed and patient may enroll if hypercalcemia returns to normal range with standard treatment).
  8. Left ventricular ejection fraction (LVEF) ≥ institutional lower limit of normal as measured by multigated acquisition scan (MUGA) scan or 2-dimensional echocardiography (ECHO) within 28 days prior to start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG).
  9. Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test prior to initiation of the SL-401 Run in Cycle (if required) and repeated with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting Pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control, 1 highly effective method and 1 additional effective method at the same time, at least 28 days before she starts taking Pomalidomide through 30 days after the last dose of Pomalidomide and 60 days after the last dose of SL-401. FCBP must also agree to ongoing pregnancy testing during the entire duration of treatment. Men must agree to use a latex or synthetic condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 60 days after the last dose of Pomalidomide or SL-401. These same patients must not donate sperm. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. All patients enrolled into this study, must agree to be registered in and must comply with all requirements of the Pomalidomide REMS(TM) program.

     * An FCBP is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

Patients will be ineligible for this study if they meet any 1 of the following criteria:

1. The patient has an active malignancy and/or cancer history that may confound the assessment of the study endpoints. Patients with a past cancer history (within 2 years of entry) with substantial potential for recurrence and/or ongoing active malignancy must be discussed with the Sponsor before study entry. Patients with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including superficial bladder cancer), cervical intraepithelial neoplasia, organ-confined prostate cancer with no evidence of progressive disease.
2. Prior therapy with SL-401 or received any investigational drug within the prior 30 days or 5 half-lives of the investigational drug, whichever is longer.
3. Prior anti-cancer therapy (chemotherapy, targeted agents, radiotherapy, and immunotherapy) within the prior 14 days except for alkylating agents (e.g., melphalan) within the prior 28 days.
4. Pomalidomide (POM)-refractory disease (i.e., non-responsive to prior POM [either as monotherapy or in combination] or relapse/progressive disease within 60 days of prior POM (either as monotherapy or in combination). Prior POM exposure is permitted, provided the patient's MM is not considered POM-refractory as defined above.
5. Primary refractory MM defined as disease that is non-responsive in patients that have never achieved at least stable disease or better with any therapy.
6. Any > grade 1 (according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], v.4.03) adverse reaction unresolved from previous treatments or not readily managed and controlled with supportive care. The presence of alopecia of any grade and peripheral neuropathy ≤ grade 2 without pain is allowed.
7. Previous allogeneic stem cell transplantation with active graft-versus-host-disease, or treatment with immunosuppressive therapy in the 2 months prior to study entry.
8. Daily requirement for corticosteroids >10 mg prednisone daily (or equivalent); inhaled corticosteroids are permitted.
9. Patient is known to be human immunodeficiency virus positive, or have chronic or active hepatitis B (core- or surface antigen-positive) or active hepatitis C infection.
10. Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association [NYHA] Class 3 or 4, congestive heart failure, uncontrolled or unstable angina, history of myocardial infarction or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
11. Uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
12. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
13. History of erythema multiforme or severe hypersensitivity to prior Immunomodulatory Drugs (IMiDs) such as thalidomide and lenalidomide.
14. The patient is receiving medications that are strong inhibitors of CYP1A2. Patients should have discontinued strong CYP1A2 inhibitors (e.g., ciprofloxacin and fluvoxamine) at least 5 half-lives before beginning study drug.
15. The patient continues to smoke cigarettes, which can induce CYP1A2.
16. Inability to tolerate thromboprophylaxis.
17. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Dana Farber Cancer Institue, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Background] Agarwal A, Ghobrial IM. Monoclonal gammopathy of undetermined significance and smoldering multiple myeloma: a review of the current understanding of epidemiology, biology, risk stratification, and management of myeloma precursor disease. Clin Cancer Res. 2013 Mar 1;19(5):985-94. doi: 10.1158/1078-0432.CCR-12-2922. Epub 2012 Dec 5. PMID 23224402
- [Background] Aldinucci D, Olivo K, Lorenzon D, Poletto D, Gloghini A, Carbone A, Pinto A. The role of interleukin-3 in classical Hodgkin's disease. Leuk Lymphoma. 2005 Mar;46(3):303-11. doi: 10.1080/10428190400013712. PMID 15621820
- [Background] Aldinucci D, Poletto D, Gloghini A, Nanni P, Degan M, Perin T, Ceolin P, Rossi FM, Gattei V, Carbone A, Pinto A. Expression of functional interleukin-3 receptors on Hodgkin and Reed-Sternberg cells. Am J Pathol. 2002 Feb;160(2):585-96. doi: 10.1016/S0002-9440(10)64878-X. PMID 11839579
- [Background] Alexander RL, Kucera GL, Klein B, Frankel AE. In vitro interleukin-3 binding to leukemia cells predicts cytotoxicity of a diphtheria toxin/IL-3 fusion protein. Bioconjug Chem. 2000 Jul-Aug;11(4):564-8. doi: 10.1021/bc000009q. PMID 10898579
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Angelot-Delettre F, Frankel AE, Liu SE et al. The IL-3Rα-Targeted Drug SL-401 Selectively kills Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) Cells. ASH 2011, Poster #2588.
- [Background] Bao S, Wu Q, McLendon RE, Hao Y, Shi Q, Hjelmeland AB, Dewhirst MW, Bigner DD, Rich JN. Glioma stem cells promote radioresistance by preferential activation of the DNA damage response. Nature. 2006 Dec 7;444(7120):756-60. doi: 10.1038/nature05236. Epub 2006 Oct 18. PMID 17051156
- [Background] Black JH, McCubrey JA, Willingham MC, Ramage J, Hogge DE, Frankel AE. Diphtheria toxin-interleukin-3 fusion protein (DT(388)IL3) prolongs disease-free survival of leukemic immunocompromised mice. Leukemia. 2003 Jan;17(1):155-9. doi: 10.1038/sj.leu.2402744. PMID 12529673
- [Background] Chauhan D, Ray A, Brooks C et al. A Novel Agent SL-401 Targeting Interleukin-3 (IL-3)- Receptor Blocks Plasmacytoid Dendritic Cell (pDC)-induced Myeloma Cell Growth and Overcomes Drug Resistance. J Clin Oncol 2013; 31;(suppl; abstr 8582).
- [Background] Chauhan D, Singh AV, Brahmandam M, Carrasco R, Bandi M, Hideshima T, Bianchi G, Podar K, Tai YT, Mitsiades C, Raje N, Jaye DL, Kumar SK, Richardson P, Munshi N, Anderson KC. Functional interaction of plasmacytoid dendritic cells with multiple myeloma cells: a therapeutic target. Cancer Cell. 2009 Oct 6;16(4):309-23. doi: 10.1016/j.ccr.2009.08.019. PMID 19800576
- [Background] Chauhan D, Uchiyama H, Akbarali Y, Urashima M, Yamamoto K, Libermann TA, Anderson KC. Multiple myeloma cell adhesion-induced interleukin-6 expression in bone marrow stromal cells involves activation of NF-kappa B. Blood. 1996 Feb 1;87(3):1104-12. PMID 8562936
- [Background] Deng Q, Barbieri JT. Molecular mechanisms of the cytotoxicity of ADP-ribosylating toxins. Annu Rev Microbiol. 2008;62:271-88. doi: 10.1146/annurev.micro.62.081307.162848. PMID 18785839
- [Background] Feuring-Buske M, Frankel AE, Alexander RL, Gerhard B, Hogge DE. A diphtheria toxin-interleukin 3 fusion protein is cytotoxic to primitive acute myeloid leukemia progenitors but spares normal progenitors. Cancer Res. 2002 Mar 15;62(6):1730-6. PMID 11912147
- [Background] FitzGerald D, Pastan I. Targeted toxin therapy for the treatment of cancer. J Natl Cancer Inst. 1989 Oct 4;81(19):1455-63. doi: 10.1093/jnci/81.19.1455. PMID 2550658
- [Background] Florian S, Sonneck K, Hauswirth AW, Krauth MT, Schernthaner GH, Sperr WR, Valent P. Detection of molecular targets on the surface of CD34+/CD38-- stem cells in various myeloid malignancies. Leuk Lymphoma. 2006 Feb;47(2):207-22. doi: 10.1080/10428190500272507. PMID 16321850
- [Background] Frankel AE, McCubrey JA, Miller MS, Delatte S, Ramage J, Kiser M, Kucera GL, Alexander RL, Beran M, Tagge EP, Kreitman RJ, Hogge DE. Diphtheria toxin fused to human interleukin-3 is toxic to blasts from patients with myeloid leukemias. Leukemia. 2000 Apr;14(4):576-85. doi: 10.1038/sj.leu.2401743. PMID 10764142
- [Background] Frolova O, Frankel AE, Korchin B et al. IL3R-Directed Agents, SL-401 and SL-501, Inhibit the Growth of Leukemia Stem cells in CML. Blood (ASH Meeting Abstracts) 2010 116: Abstract 3403.
- [Background] Giles F, O'Brien S, Cortes J, Verstovsek S, Bueso-Ramos C, Shan J, Pierce S, Garcia-Manero G, Keating M, Kantarjian H. Outcome of patients with acute myelogenous leukemia after second salvage therapy. Cancer. 2005 Aug 1;104(3):547-54. doi: 10.1002/cncr.21187. PMID 15973664
- [Background] Hermann PC, Huber SL, Heeschen C. Metastatic cancer stem cells: a new target for anti-cancer therapy? Cell Cycle. 2008 Jan 15;7(2):188-93. doi: 10.4161/cc.7.2.5326. Epub 2007 Nov 18. PMID 18256530
- [Background] Jordan CT, Guzman ML, Noble M. Cancer stem cells. N Engl J Med. 2006 Sep 21;355(12):1253-61. doi: 10.1056/NEJMra061808. No abstract available. PMID 16990388
- [Background] Jordan CT, Upchurch D, Szilvassy SJ, Guzman ML, Howard DS, Pettigrew AL, Meyerrose T, Rossi R, Grimes B, Rizzieri DA, Luger SM, Phillips GL. The interleukin-3 receptor alpha chain is a unique marker for human acute myelogenous leukemia stem cells. Leukemia. 2000 Oct;14(10):1777-84. doi: 10.1038/sj.leu.2401903. PMID 11021753
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Lhermitte L, de Labarthe A, Dupret C, Lapillonne H, Millien C, Landman-Parker J, Hermine O, Baruchel A, Sigaux F, Macintyre E, Asnafi V. Most immature T-ALLs express Ra-IL3 (CD123): possible target for DT-IL3 therapy. Leukemia. 2006 Oct;20(10):1908-10. doi: 10.1038/sj.leu.2404349. Epub 2006 Aug 10. No abstract available. PMID 16900212
- [Background] Louie GV, Yang W, Bowman ME, Choe S. Crystal structure of the complex of diphtheria toxin with an extracellular fragment of its receptor. Mol Cell. 1997 Dec;1(1):67-78. doi: 10.1016/s1097-2765(00)80008-8. PMID 9659904
- [Background] McCann S, Akilov OE, Geskin L. Adverse effects of denileukin diftitox and their management in patients with cutaneous T-cell lymphoma. Clin J Oncol Nurs. 2012 Oct;16(5):E164-72. doi: 10.1188/12.CJON.E164-E172. PMID 23022942
- [Background] Munoz L, Nomdedeu JF, Lopez O, Carnicer MJ, Bellido M, Aventin A, Brunet S, Sierra J. Interleukin-3 receptor alpha chain (CD123) is widely expressed in hematologic malignancies. Haematologica. 2001 Dec;86(12):1261-9. PMID 11726317
- [Background] National Cancer Institute-Common Terminology Criteria: Version 4.03 reference, accessible through the NCI website at http://ctep.info.nih.gov/reporting/ctc.html.
- [Background] Olsen E, Duvic M, Frankel A, Kim Y, Martin A, Vonderheid E, Jegasothy B, Wood G, Gordon M, Heald P, Oseroff A, Pinter-Brown L, Bowen G, Kuzel T, Fivenson D, Foss F, Glode M, Molina A, Knobler E, Stewart S, Cooper K, Stevens S, Craig F, Reuben J, Bacha P, Nichols J. Pivotal phase III trial of two dose levels of denileukin diftitox for the treatment of cutaneous T-cell lymphoma. J Clin Oncol. 2001 Jan 15;19(2):376-88. doi: 10.1200/JCO.2001.19.2.376. PMID 11208829
- [Background] Perentesis JP, Miller SP, Bodley JW. Protein toxin inhibitors of protein synthesis. Biofactors. 1992 Jan;3(3):173-84. PMID 1599611
- [Background] Pomalidomide Perscribing Information. POMPI.001/MG.001 02/13. Reference ID: 325852
- [Background] Prince HM, Duvic M, Martin A, Sterry W, Assaf C, Sun Y, Straus D, Acosta M, Negro-Vilar A. Phase III placebo-controlled trial of denileukin diftitox for patients with cutaneous T-cell lymphoma. J Clin Oncol. 2010 Apr 10;28(11):1870-7. doi: 10.1200/JCO.2009.26.2386. Epub 2010 Mar 8. PMID 20212249
- [Background] Ratts R, Trujillo C, Bharti A, vanderSpek J, Harrison R, Murphy JR. A conserved motif in transmembrane helix 1 of diphtheria toxin mediates catalytic domain delivery to the cytosol. Proc Natl Acad Sci U S A. 2005 Oct 25;102(43):15635-40. doi: 10.1073/pnas.0504937102. Epub 2005 Oct 17. PMID 16230620
- [Background] Richardson PG, Siegel DS, Vij R, Hofmeister CC, Baz R, Jagannath S, Chen C, Lonial S, Jakubowiak A, Bahlis N, Song K, Belch A, Raje N, Shustik C, Lentzsch S, Lacy M, Mikhael J, Matous J, Vesole D, Chen M, Zaki MH, Jacques C, Yu Z, Anderson KC. Pomalidomide alone or in combination with low-dose dexamethasone in relapsed and refractory multiple myeloma: a randomized phase 2 study. Blood. 2014 Mar 20;123(12):1826-32. doi: 10.1182/blood-2013-11-538835. Epub 2014 Jan 13. PMID 24421329
- [Background] Miguel JS, Weisel K, Moreau P, Lacy M, Song K, Delforge M, Karlin L, Goldschmidt H, Banos A, Oriol A, Alegre A, Chen C, Cavo M, Garderet L, Ivanova V, Martinez-Lopez J, Belch A, Palumbo A, Schey S, Sonneveld P, Yu X, Sternas L, Jacques C, Zaki M, Dimopoulos M. Pomalidomide plus low-dose dexamethasone versus high-dose dexamethasone alone for patients with relapsed and refractory multiple myeloma (MM-003): a randomised, open-label, phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1055-1066. doi: 10.1016/S1470-2045(13)70380-2. Epub 2013 Sep 3. PMID 24007748
- [Background] Tehranchi R, Woll PS, Anderson K, Buza-Vidas N, Mizukami T, Mead AJ, Astrand-Grundstrom I, Strombeck B, Horvat A, Ferry H, Dhanda RS, Hast R, Ryden T, Vyas P, Gohring G, Schlegelberger B, Johansson B, Hellstrom-Lindberg E, List A, Nilsson L, Jacobsen SE. Persistent malignant stem cells in del(5q) myelodysplasia in remission. N Engl J Med. 2010 Sep 9;363(11):1025-37. doi: 10.1056/NEJMoa0912228. PMID 20825315
- [Background] Thorburn A, Thorburn J, Frankel AE. Induction of apoptosis by tumor cell-targeted toxins. Apoptosis. 2004 Jan;9(1):19-25. doi: 10.1023/B:APPT.0000012118.95548.88. PMID 14739595
- [Background] van Rhenen A, Feller N, Kelder A, Westra AH, Rombouts E, Zweegman S, van der Pol MA, Waisfisz Q, Ossenkoppele GJ, Schuurhuis GJ. High stem cell frequency in acute myeloid leukemia at diagnosis predicts high minimal residual disease and poor survival. Clin Cancer Res. 2005 Sep 15;11(18):6520-7. doi: 10.1158/1078-0432.CCR-05-0468. PMID 16166428
- [Background] Vergez F, Green AS, Tamburini J, Sarry JE, Gaillard B, Cornillet-Lefebvre P, Pannetier M, Neyret A, Chapuis N, Ifrah N, Dreyfus F, Manenti S, Demur C, Delabesse E, Lacombe C, Mayeux P, Bouscary D, Recher C, Bardet V. High levels of CD34+CD38low/-CD123+ blasts are predictive of an adverse outcome in acute myeloid leukemia: a Groupe Ouest-Est des Leucemies Aigues et Maladies du Sang (GOELAMS) study. Haematologica. 2011 Dec;96(12):1792-8. doi: 10.3324/haematol.2011.047894. Epub 2011 Sep 20. PMID 21933861
- [Background] Yamaizumi M, Mekada E, Uchida T, Okada Y. One molecule of diphtheria toxin fragment A introduced into a cell can kill the cell. Cell. 1978 Sep;15(1):245-50. doi: 10.1016/0092-8674(78)90099-5. PMID 699044
- [Background] Zeppernick F, Ahmadi R, Campos B, Dictus C, Helmke BM, Becker N, Lichter P, Unterberg A, Radlwimmer B, Herold-Mende CC. Stem cell marker CD133 affects clinical outcome in glioma patients. Clin Cancer Res. 2008 Jan 1;14(1):123-9. doi: 10.1158/1078-0432.CCR-07-0932. PMID 18172261

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, SL-401 7 µg/kg/Day: Phase 1, SL-401 7 µg/kg/day in combination with Pomalidomide and Dexamethasone
- Phase 1, SL-401 9 µg/kg/Day: Phase 1, SL-401 9 µg/kg/day in combination with Pomalidomide and Dexamethasone
Period: Overall Study
Arm/Group | Phase 1, SL-401 7 µg/kg/Day | Phase 1, SL-401 9 µg/kg/Day
Started | 7 | 2
Completed | 0 | 0
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive Disease | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- SL-401 7 µg/kg/Day: SL-401 7 µg/kg/day in combination with Pomalidomide and Dexamethasone
  SL-401 7 µg/kg/day: SL-401 7 µg/kg/day in combination with Pomalidomide/Dexamethasone
- SL-401 9 µg/kg/Day: SL-401 9 µg/kg/day in combination with Pomalidomide and Dexamethasone
  SL-401 9 µg/kg/day: SL-401 9 µg/kg/day in combination with Pomalidomide/Dexamethasone
- Total: Total of all reporting groups
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (4.35) | 57.0 (0.00) | 63.4 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9
Height [Mean (Standard Deviation); unit: cm] | 164.6 (14.39) | 164.7 (6.65) | 164.6 (12.42)
Weight [Mean (Standard Deviation); unit: kg] | 85.6 (18.40) | 92.9 (16.62) | 87.2 (17.29)
Eastern Cooperative Oncology Group Status (ECOG Status) [Count of Participants; unit: Participants] — ECOG Performance Status Scale 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 3 | 2 | 5
    1 | 4 | 0 | 4
    2 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicities and Treatment-emergent Adverse Events
Description: To evaluate the safety of single agent SL-401 in an initial run-in cycle in patients with multiple myeloma
Time Frame: For a 28-day cycle, Cycle 1
Measure: Count of Participants; unit: Participants
Groups:
- SL-401 7 µg/kg/Day: SL-401 7 µg/kg/day in combination with pomalidomide and dexamethasone
- SL-401 9 µg/kg/Day: SL-401 9 µg/kg/day in combination with pomalidomide and dexamethasone
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
Number analyzed (Participants) | 7 | 2
Participants | 7 | 2

2. Primary Outcome: Number of Patients With Treatment-related Adverse Events
Description: To evaluate the safety of single agent SL-401 in an initial run-in cycle in patients with multiple myeloma
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
Number analyzed (Participants) | 7 | 2
Participants
  At Least 1 Treatment-Related Treatment-Emergent Adverse Event | 7 | 2
  Fatigue | 5 | 1
  Nausea | 5 | 1
  Pyrexia | 4 | 2
  Hypoalbuminaemia | 4 | 1
  Chills | 4 | 0
  Insomnia | 3 | 1
  Aspartate aminotransferase increased | 2 | 1
  Constipation | 2 | 1
  Dizziness | 3 | 0
  Flushing | 3 | 0
  Headache | 2 | 1
  Hypophosphataemia | 2 | 1
  Neutropenia | 3 | 0
  Oedema peripheral | 3 | 0
  Thrombocytopenia | 2 | 1

3. Primary Outcome: Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug
Description: To evaluate the safety of single agent SL-401 in an initial run-in cycle in patients with multiple myeloma (MM)
Time Frame: Up to 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- SL-401 7 µg/kg/Day: SL-401 7 µg/kg/day in combination with pomalidomide/dexamethasone (pom/dex)
  SL-401 7 µg/kg/day: SL-401 7 µg/kg/day in combination with pomalidomide/dexamethasone (pom/dex)
- SL-401 9 µg/kg/Day: SL-401 9 µg/kg/day in combination with pomalidomide/dexamethasone (pom/dex)
  SL-401 9 µg/kg/day: SL-401 9 µg/kg/day in combination with pomalidomide/dexamethasone (pom/dex)
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
Number analyzed (Participants) | 7 | 2
Participants
  At Least 1 TEAE Leading to Discontinuation of Study Drug | 1 | 1
  Capillary leak syndrome | 0 | 1
  Metastatic malignant melanoma | 1 | 0
  Pancreatitis | 0 | 1
  Thrombocytopenia | 0 | 1

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as complete response + very good partial response + partial response and clinical benefit rate (CR + VGPR + PR + minimal response [MR]) based on International Myeloma Working Group-defined response criteria and the duration of response (DOR) in relapsed refractory multiple myeloma (RRMM) patients.
Time Frame: Up to 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
Number analyzed (Participants) | 5 | 1
Participants
  Overall Response Rate | 5 | 0
  Complete Response | 0 | 0
  Stringent Complete Response | 0 | 0
  Very Good Partial Response | 0 | 0
  Partial Response | 5 | 0
  Minimal Response | 0 | 0
  Stable Disease | 0 | 1
  Progressive Disease | 0 | 0
  Progressive Disease or Death After Overall Response | 1 | 0
  Censored | 4 | 0

5. Secondary Outcome: Progression-free Survival
Description: Per International Myeloma Working Group Response Criteria, progression/progressive disease is defined as increase of >25% from lowest response value in any 1 of the following: serum M-component (the absolute increase must be >0.5 g/dL)4 and/or urine M-component (the absolute increase must be >200 mg/24 h) and/or; only in patients without measurable serum and urine M-protein, the difference between involved and uninvolved FLC levels. The absolute increase must be >10 mg/dL; only in patients without measurable serum and urine M-protein and without measurable disease by FLC levels; bone marrow plasma cell percentage (absolute % must be ≥10%); definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: Up to 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
Number analyzed (Participants) | 5 | 1
Participants
  Disease Progression | 1 | 0
  Death | 0 | 0
  Censored | 4 | 1
  PFS at 6 Months | 4 | 0
  PFS at 12 Months | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SL-401 7 µg/kg/Day | SL-401 9 µg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/7 | 2/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SL-401 7 µg/kg/Day (N=7) | SL-401 9 µg/kg/Day (N=2)
Pneumonia (Infections and infestations) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SL-401 7 µg/kg/Day (N=7) | SL-401 9 µg/kg/Day (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Hypermetropia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 5 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 2
Malaise (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
C-reactive protein increased (Investigations) | 0 | 1
Glucose urine (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Emotional distress (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow accrual and changes to Sponsor's development program priorities. The third dose level (12 µg/kg/day), for Phase 2, was not investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution's individual results may be submitted for publication only after the results of the multicenter study are published, 18 months after study completion at all sites, or notification from Stemline Therapeutics, Inc. that submission of a multicenter publication is no longer planned, whichever shall occur first.

DOCUMENTS (2):
  • Study Protocol (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02661022/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT02661022/SAP_001.pdf